CLINICAL TRIAL: NCT00572013
Title: A Phase I/II Trial of Rituxan and BEAM High-Dose Chemotherapy and Autologous Peripheral Blood Progenitor Transplant for Indolent Lymphoma
Brief Title: Rituxan and BEAM With Autologous Peripheral Blood Progenitor Transplant for Indolent Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0138-98-FB
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I Rituxan and BEAM post-autologous stem cell transplant (Experimental): Rituxan and BEAM [Carmustine (BCNU), Etoposide, Cytarabine (Ara-C, cytosine arabinoside), Melphalan] will be a pre- and post-transplant agent to aid in the chemotherapy sensitization post-autologous stem cell transplant.
  Interventions: Drug: Rituxan; Drug: BEAM; Procedure: Autologous stem cell transplant

INTERVENTIONS:
Drug: Rituxan — 375mg/m2 IV on days -20 to -8. Infusion to begin at rate of 50mg/hour for 1st hour.If no toxicity rate may be increased. A second infusion 375mg/m2 given 30days post transplant and again at 60 days post transplant
  Other Names: Rituximab
Drug: BEAM — BCNU(carmustine)on day -6 300mg/M2 IV, etoposide 100mg/M2 BID on days -5 through -2, cytarabine 100mg/m2 BID on days -5 through -2, melphalan 140mg/m2 IV on day -1
Procedure: Autologous stem cell transplant — following chemotherapy, on day 0 of treatment, the previously stored hematopoietic stem cells will be reinfused via the central venous line

SUMMARY:
To determine the response rate, complete and partial, of patients with indolent lymphoma receiving Rituxan and BEAM with autologous stem cell transplant.

DETAILED DESCRIPTION:
Objectives: I. To determine the response rate, complete and partial, of patients with indolent lymphoma receiving Rituxan and BEAM with autologous stem cell transplant. II. To determine if the addition of Rituxan changes the toxicity profile attributed to high-dose BEAM chemotherapy.

This protocol is a phase I/II trial combining the Rituxan as a pre and post-transplant agent to aid in the chemotherapy sensitization and the treatment of minimal residual disease post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Any low-grade B-cell, CD20 positive, non-Hodgkin's lymphoma that is felt to otherwise be a transplant candidate (relapsed, induction failure, first PR or CR).

  o Small lymphocytic, marginal zone, mantle cell, and follicular histologies.
* At least 19 years of age
* Signed written informed consent
* Expected survival of at least 6 months
* WHO performance status greater or equal to 2
* Male or female subjects of reproductive potential who are able to follow accepted birth control measures.

Exclusion Criteria:

* No history of T-cell lymphoma
* Not pregnant or lactating women
* No serious disease or condition that, in the opinion of the investigator, would compromise the subject's ability to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1998-05-12 (Actual); Primary Completion 2001-01-01 (Actual); Study Completion 2009-09-18 (Actual)

PRIMARY OUTCOMES:
Response rate | 100 day
  Disease response at day 100

SECONDARY OUTCOMES:
Overall survival | diagnosis until death
  Survival time from diagnosis until death

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Section of Oncology/Hematology, Omaha, Nebraska, United States